CLINICAL TRIAL: NCT04957849
Title: The Neuroendoscopic, Trans-occipital Approach Evacuation of Acute Hypertensive Cerebral Hemmorrhage Combined Low-drainage Surgery: a Multi-center Clinical Trial
Brief Title: Acute Hypertensive Cerebral Hemmorrhage Surgery
Acronym: NET-OCEAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Huashan Hospital (Other); Tianjin Medical University General Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Peking Union Medical College Hospital (Other); Second Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital of Nanchang University (Other); The General Hospital of Eastern Theater Command (Other); First Affiliated Hospital of Harbin Medical University (Other); Shengjing Hospital (Other); ShuGuang Hospital (Other); Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Hou Lijun, Professor, Shanghai Changzheng Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NET-OCEAN
Record Dates: First submitted 2021-07-03; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Hypertensive Intracerebral Hemorrhage
Keywords: neuroendoscope; trans-occipital approach; Acute Hypertensive Cerebral Hemmorrhage; Low-drainage Surgery
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-frontal keyhole approach (Active Comparator): After general anesthesia, the patient was placed in supine position with head frame fixed. A straight or arc incision was made in the hairline of the affected side. The incision was 3cm beside the midline. The length of the incision was about 4cm and the diameter of the bone window was about 2.5cm. According to the preoperative thin-layer CT scan, the dura mater and part of the cerebral cortex were cut, and the endoport and other hard channels were inserted. The incision reached 2 / 3 of the length of the hematoma along the direction parallel to the long axis of the hematoma, During the operation, mini aneurysms were clipped to close the responsible vessels, and hemostatic gauze was applied on the surface of the hematoma cavity. Silica gel external drainage tube was placed in the hematoma cavity. The external drainage tube led out the skin through the subcutaneous tunnel, and the dura was sutured.
  Interventions: Procedure: Endoscopic Evacuation of Acute Hypertensive Intracerebral Hemorrhage via Trans-frontal keyhole approach
- Trans-occipital keyhole approach (Active Comparator): After general anesthesia, the patient was placed in prone position with head frame fixed. According to the preoperative thin-layer CT scan, the long axis of hematoma was perpendicular to the ground, and the occipital puncture point was found along the extension line of the long axis of hematoma. Taking the puncture point as the center, a straight or arc incision parallel to the sagittal sinus was taken. The length of the incision was about 4cm, and the diameter of the bone window was about 2.5cm, Endoport and other hard channels were inserted to reach 2 / 3 of the long diameter of the hematoma along the direction parallel to the long axis of the hematoma. Under the neuroendoscope, the hematoma was aspirated or resected in blocks. During the operation, mini aneurysm clamp was used to clamp the responsible vessels, and hemostatic gauze was applied on the surface of the hematoma cavity. Silica gel external drainage tube was placed in the hematoma cavity.
  Interventions: Procedure: The Neuroendoscopic, Trans-occipital Approach Evacuation of Acute Hypertensive Cerebral Hemmorrhage Combined Low-drainage Surgery

INTERVENTIONS:
Procedure: The Neuroendoscopic, Trans-occipital Approach Evacuation of Acute Hypertensive Cerebral Hemmorrhage Combined Low-drainage Surgery — The Neuroendoscopic, Trans-occipital Approach Evacuation of Acute Hypertensive Cerebral Hemmorrhage Combined Low-drainage Surgery
  Arms: Trans-occipital keyhole approach
Procedure: Endoscopic Evacuation of Acute Hypertensive Intracerebral Hemorrhage via Trans-frontal keyhole approach — Endoscopic Evacuation of Acute Hypertensive Intracerebral Hemorrhage via Trans-frontal keyhole approach
  Arms: Trans-frontal keyhole approach

SUMMARY:
The Neuroendoscopic, Trans-occipital Approach Evacuation of Acute Hypertensive Cerebral Hemmorrhage Combined Low-drainage Surgery: a Multi-center Clinical Trial

DETAILED DESCRIPTION:
To evaluate the effect of different surgical approaches on the prognosis of patients with hypertensive intracerebral hemorrhage, hypertensive patients who met the diagnostic criteria of American guidelines for the treatment of adult spontaneous intracerebral hemorrhage (2015) were selected. The time from onset to admission was less than 8 hours. Blood routine examination, liver and kidney function, coagulation system, infectious diseases and other examinations were performed before operation, with emergency surgical indications, They were divided into two groups: transfrontal keyhole approach and transoccipital keyhole approach. Emergency endoscopic hematoma removal was performed. The patients were systematically evaluated and followed up at 1 week, 1 month, 3 months, 6 months and 12 months after operation to observe the improvement of consciousness, GCS score, postoperative rebleeding (appearance, bleeding volume, location, broken into ventricle, etc.), The prognosis was evaluated by ADL score, GCS score, gos score, modified Rankin scale, Mrs scale and ICH Score (GCS, hematoma volume, intraventricular hemorrhage, infratentorial source, patient age, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed patients with spontaneous cerebral hemorrhage in the basal ganglia (in line with the diagnostic criteria of the American Adult Spontaneous Cerebral Hemorrhage Treatment Guidelines (2015)).
2. Head CT showed; hematoma volume ≥ 30ml, intraventricular hemorrhage is not counted as hemorrhage volume.
3. Time from onset to hospital admission ≤8h.
4. The age of the patient is 15-75 years old.
5. Glasgow Coma Score (GCS)> 5 points.
6. The patient/family knows and signs the informed consent form.
7. Have a clear history of hypertension in the past.

Exclusion Criteria:

1. Bleeding caused by aneurysm, vascular malformation or tumor stroke.
2. Combined with a history of head injury or trauma.
3. There is more blood in the skull.
4. Past mental disorders or neurological dysfunction.
5. A history of procoagulant dysfunction or anticoagulant drugs.
6. Patients with complications such as liver and kidney dysfunction.
7. Those with poor compliance.
8. Pregnant patients.
9. With massive hemorrhage of the ventricle (the area of the hematoma in the CT side is larger than 1/2 of the transverse section), hemorrhage in the third and fourth ventricles with enlarged ventricles.
10. With late-stage cerebral herniation (bilateral dilated pupils, central respiratory and circulatory failure).
11. Severe cardiovascular and cerebrovascular diseases: such as myocardial infarction, cerebral infarction, coronary heart disease, myocarditis, malignant arrhythmia, etc.
12. Participate in other clinical research 3 months before enrollment.
13. The doctor in charge believes that the study plan cannot be followed.
14. Those who are or plan to become pregnant or breastfeeding.
15. Those who are known to be allergic to test drugs or related products.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate | 1 month postoperation
  The evaluation criteria of complete remission: more than 85% of intracranial hematoma was cleared, mild brain edema, and the postoperative hospital stay was less than 2 weeks. The evaluation criteria of partial remission: the clearance rate of intracranial hematoma was 60% - 85%, the postoperative brain edema was obvious, and the postoperative hospital stay was less than 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Hou, MD,PhD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Department of Neurosurgery, Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No